CLINICAL TRIAL: NCT05167643
Title: Exploratory Study of HR-positive HER2-positive MBC Combined Treatment Plan
Brief Title: H (Trastuzumab or Biosimilar) Combined With CDK4/6 Inhibitor + AI±OFS in the Treatment of HR+HER2+ Advanced Breast Cancer Efficacy and Safety: a Chinese Multi-center Real World Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BC-CIH-H-RWS
Record Dates: First submitted 2021-11-03; First posted 2021-12-22 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2021-10

CONDITIONS: Advanced HR+ HER2 Negative Breast Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trastuzumab injection+Piperacillil tablets+Letrozole tablets (Experimental): Trastuzumab injection:Once in 21 days IVD；Piperacillil tablets:125mg qd (d1-21) PO；Letrozole tablets:2.5mg POqd；According to the current clinical guidelines combined with clinical practice, the treating physicians recommended the treatment plan to the subjects, and decided to enroll HR+/HER2+ advanced breast cancer patients treated with H combined with CDK4/6 inhibitor + AI±OFS into this study
  Interventions: Drug: Enituzumab injection+Abesili tablets+Anastrozole tablets

INTERVENTIONS:
Drug: Enituzumab injection+Abesili tablets+Anastrozole tablets — According to the current clinical guidelines combined with clinical practice, the treating physicians recommended the treatment plan to the subjects, and decided to enroll HR+/HER2+ advanced breast cancer patients treated with H combined with CDK4/6 inhibitor + AI±OFS into this study

SUMMARY:
This study is a multi-center prospective real-world clinical study, mainly evaluating the efficacy and safety of H combined with CDK4/6 inhibitor + AI in the treatment of HR+/HER2+ advanced breast cancer; exploring potential biomarkers.

DETAILED DESCRIPTION:
This study is a multi-center, prospective. Because of the non-interventional nature of this study, the choice of H can be trastuzumab, biosimilar drugs Hantriyou, enituzumab, etc. The CDK4/6 inhibitor can be piperazil, abecilil and the like. AI can be letrozole, anastrozole, exemestane. This study does not change or interfere with clinicians' diagnosis and treatment decisions, as well as patients' actual medical practices.This real-world study will not do formal inference statistical analysis. All hypothesis testing is exploratory. A comprehensive statistical analysis plan (SAP) will be prepared and finalized before the data is locked and analyzed. Descriptive statistics will be performed, including the number and percentage of categorical variables, as well as the number, average, standard deviation, median, maximum, and minimum of continuous variables. Kaplan-Meier survival analysis was used to calculate the median PFS and OS and their 95% confidence intervals. The median time to disease progression and median survival time will also be calculated, as well as its 95% confidence interval. ORR and CBR will be analyzed and expressed by the ratio and the corresponding 95% confidence interval (CI). The multivariate logistic regression model was used to calculate the odds ratio (OR) and its 95% confidence interval and p-value. The subgroup analysis of PFS and OS was analyzed by Log-rank test. The COX proportional hazard regression model is used to calculate the hazard ratio and its 95% confidence interval.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old.
2. HR-positive and HER2-positive breast cancer diagnosed pathologically.

   1. ER positive and/or PR positive is defined as: the proportion of positively stained tumor cells in all tumor cells is ≥10% (reviewed and confirmed by the investigator at the test center);
   2. HER2 positive is defined as: standard immunohistochemistry (IHC) test for HER2 (3+), or HER2 (2+), FISH test is positive (reviewed and confirmed by the investigator at the test center).
3. After H-based combined chemotherapy treatment has progressed (≤1 line), or the combined treatment is effective but not suitable for continued combined chemotherapy; or initially unsuitable for targeted combined chemotherapy for recurrent metastatic breast cancer or inoperable locally advanced breast cancer Breast cancer patients.
4. Postmenopausal or premenopausal/perimenopausal female patients can be included in the group. Premenopausal or perimenopausal female patients must be willing to receive LHRHa treatment during the study period.
5. According to the RECIST 1.1 standard, patients can have: a) measurable lesions; b) without measurable lesions, unmeasurable osteolytic or mixed (osteolytic + osteogenic) bone lesions. c) Unmeasurable lesions.
6. The main organs are functioning normally, that is, they meet the following standards:

   1. The standard of routine blood examination should meet:

      Hb≥80 g/L; ANC≥1.5×109 /L; PLT≥75×109 /L;
   2. The biochemical inspection shall meet the following standards:

      TBIL≤1.5×ULN (upper limit of normal value); ALT and AST≤2.5×ULN; if there is liver metastasis, ALT and AST≤5×ULN; Serum creatinine ≤1.5×ULN, creatinine clearance ≥50ml/min (based on Cockroft and Gault formula);
   3. Heart color Doppler ultrasound Left ventricular ejection fraction (LVEF) ≥50%.

Exclusion Criteria:

1. Patients who have previously received CDK4/6 inhibitor drug therapy.
2. T-DM1 treats patients.
3. Female patients during pregnancy or lactation.
4. Suffer from serious concomitant diseases, such as infectious diseases; there are many factors that affect the oral and absorption of drugs.
5. Patients considered by the investigator to be unsuitable to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-01-23 (Actual); Primary Completion 2022-10-23 (Estimated); Study Completion 2024-08-23 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Estimated 24 months
  From enrollment to progression or death (for any reason)

SECONDARY OUTCOMES:
Objective response rate (ORR) | Estimated 24 months
  Ratio of CR and PR in all subjects
Disease Control Rate (DCR) | Estimated 24 months
  Ratio of CR ,PR and SD in all subjects
Overall survival (OS) | Estimated 36 months
  From enrollment to death (for any reason)
Security (CTCAE 5.0) | From informed consent through 28 days following treatment completion
  Adverse events are described in terms of CTCAE 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Chunfang Hao, PhD, Principal Investigator — Department of Breast Cancer Medical Oncology
Locations (1):
- Tianjin Cancer Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: No